CLINICAL TRIAL: NCT01255592
Title: A Phase II Randomised, Double-Blind, Placebo-Controlled, Parallel Group Study to Assess the Efficacy of 28-Day Oral Administration of AZD5069 Twice Daily in Patients With Bronchiectasis
Brief Title: Evaluation of the Effect of AZD5069 in Patients With Bronchiectasis
Acronym: STRATUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3550C00014
Record Dates: First submitted 2010-12-02; First posted 2010-12-07 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Bronchiectasis; Lung Disease; Respiratory Diseases
Keywords: Bronchiectasis; Neutrophil; Respiratory disease; Sputum
MeSH Terms: conditions — Bronchiectasis; Lung Diseases; Respiratory Tract Diseases; Respiration Disorders | interventions — N-(2-(2,3-difluoro-6-benzylthio)-6-(3,4-dihydroxybutan-2-yloxy)pyrimidin-4-yl)azetidine-1-sulfonamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Treatment arm AZD5069
  Interventions: Drug: AZD5069
- 2 (Placebo Comparator): Placebo dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5069 — Oral dose bid
  Arms: 1
Drug: Placebo — Oral dose bid
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the effect of AZD5069 in patients with bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* Male, or female of non-child bearing potential; ie, women who are permanently or surgically sterilised or post-menopausal.
* Aged 18 to 80 years inclusive at screening (Visit 1)
* Have a clinical diagnosis of idiopathic or post infective bronchiectasis as diagnosed with a historical high resolution computerised tomography (HRCT) or bronchogram
* Be sputum producers with a history of chronic expectoration on most days of most weeks of the year. Patients should have a history of spontaneously producing sputum on a daily basis and should be able to provide at least 2 of the 3 required baseline sputum samples with an average of 3 mL or more.
* Be on a stable treatment regimen, as judged by the investigator.

Exclusion Criteria:

* Any clinically significant disease or disorder
* Patients with other latent or chronic infections or at risk of infection within 90 days before Visit 2
* An acute exacerbation or acute respiratory infection (upper or lower) requiring oral steroids or antibiotics within 30 days prior to Visit 2
* An FEV1 of <30% of predicted normal at Visit 1
* Patients who have received live or live-attenuated vaccine in the 2 weeks prior to dosing (Visit 2)
* Concomitant diagnosis of significant pulmonary disease other than bronchiectasis or COPD, including symptomatic asthma and allergic bronchopulmonary aspergillosis
* Bronchiectasis associated with a generalised immunodeficiency disorder, where manifestations other than bronchiectasis predominate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Larsson,, M.B, Study Director — AstraZeneca R&D Mölndal
Locations (15):
- Czechia (2):
  - Research Site, Ostrava
  - Research Site, Prague
- Poland (3):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Warsaw
- United Kingdom (10):
  - Research Site, Hull, East Yorkshire
  - Research Site, Leicester, Leicestershire
  - Research Site, Birmingham, Wstmid
  - Research Site, Belfast
  - Research Site, Bristol
  - Research Site, Cambridge
  - Research Site, London
  - Research Site, Newcastle upon Tyne
  - Research Site, Salford
  - Research Site, Wolverhampton

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=209&filename=D3550C00014_Study_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in Europe between 27 December 2010 and 13 February 2012.
Groups:
- AZD5069: AZD5069 80 mg bd
- Placebo: Placebo for AZD5069, bd
Period: Overall Study
Arm/Group | AZD5069 | Placebo
Started | 26 | 26
Completed | 20 | 25
Not Completed | 6 | 1
Not completed — Adverse Event | 5 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo bd
- Total: Total of all reporting groups
Arm/Group | AZD5069 | Placebo | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (6.6) | 65 (8.8) | 65 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 10 | 14 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 26 | 26 | 52
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Absolute Neutrophil Cell Count in Sputum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: The PD analysis set comprised all patients who received at least 1 dose of study medication and for whom PD samples (absolute and percentage neutrophil cell count in sputum, sputum collection weight, inflammatory markers in sputum and serum) were available (assumed not to be affected by factors such as protocol violations).
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 19 | 24
ratio | 0.31 (165.925) [0.20 to 0.50] | 1.00 (213.281) [0.66 to 1.51]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; Analysis of covariance included treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection, and baseline as covariates. The analysis was done on log-transformed data. The results were back-transformed after the analysis on the log scale; Test type: Superiority or Other; p = 0.004, ANCOVA; Ratio of AZD5069 80 mg to placebo = 0.31, 90% CI 2-sided [0.17 to 0.59]

2. Secondary Outcome: Ratio of the Percentage Neutrophil Cell Count in Sputum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 19 | 24
ratio | 0.66 (29.746) [0.54 to 0.80] | 1.02 (56.883) [0.86 to 1.22]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.008, ANCOVA; Ratio of AZD5069 80 mg to placebo = 0.64, 90% CI 2-sided [0.49 to 0.84]

3. Secondary Outcome: Change From Baseline in Weight of 24-hour Sputum Collection
Description: Patients collected all sputum produced during a 24-hour period at baseline and Day 28.
Time Frame: Baseline and end of treatment (Day 28)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 20 | 25
grams | 3.51 (2.455) | -3.26 (2.195)
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; The 24-hour sputum weight on Visit 4 was compared between groups using ANCOVA (additive model) with treatment and inhaled corticosteroids/P. aeruginosa infection as fixed effects and baseline as a covariate; Test type: Superiority or Other; p = 0.047, ANCOVA; LS mean difference = 6.78, 90% CI 2-sided [1.22 to 12.33], Standard Error of Mean 3.298

4. Secondary Outcome: Change From Baseline in Slow Vital Capacity (SVC)
Description: Lung function tests consisted of 3 forced expiratory maneuvers in which the patient expired forcefully from total lung capacity to residual volume, recorded using a spirometer. SVC is the measure of the change in volume of gas in the lungs from complete inspiration to complete expiration.
Time Frame: Baseline to end of treatment (Day 28)
Population: The efficacy analysis set included all patients who were randomized (defined as having a randomization code recorded on the demography case report form), received at least one dose of study medication, and contributed sufficient data for at least one efficacy endpoint.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 23 | 26
liters | 0.05 (0.067) | -0.05 (0.063)
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; Analysis of covariance included treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection and baseline as covariates; Test type: Superiority or Other; p = 0.284, ANCOVA; LS mean difference = 0.10, 90% CI 2-sided [-0.05 to 0.26], Standard Error of Mean 0.092

5. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC)
Description: Lung function tests consisted of 3 forced expiratory maneuvers in which the patient expired forcefully from total lung capacity to residual volume, recorded using a spirometer. FVC is the maximum volume of air which can be exhaled or inspired during a forced maneuver.
Time Frame: Baseline to end of treatment (Day 28)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 24 | 26
liters | 0.07 (0.056) | 0.06 (0.054)
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.929, ANCOVA; LS mean difference = 0.01, 90% CI 2-sided [-0.12 to 0.14], Standard Error of Mean 0.078

6. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: Lung function tests consisted of 3 forced expiratory maneuvers in which the patient expired forcefully from total lung capacity to residual volume, recorded using a spirometer. FEV1 is the volume expired in the first second of maximal expiration after a full inspiration.
Time Frame: Baseline to end of treatment (Day 28)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 24 | 26
liters | -0.01 (0.044) | -0.01 (0.043)
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.966, ANCOVA; LS mean difference = -0.00, 90% CI 2-sided [-0.11 to 0.10], Standard Error of Mean 0.062

7. Secondary Outcome: Change From Baseline in Forced Expiratory Flow Between 25% and 75% of Forced Vital Capacity (FEF25-75)
Description: Lung function tests consisted of 3 forced expiratory maneuvers in which the patient expired forcefully from total lung capacity to residual volume, recorded using a spirometer. FEF25-75 is flow rate during the middle half of forced vital capacity (25%-75% of the total volume (FVC) exhaled).
Time Frame: Baseline to end of treatment (Day 28)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 24 | 25
liters/second | -0.04 (0.063) | -0.07 (0.062)
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.791, ANCOVA; LS mean difference = 0.02, 90% CI 2-sided [-0.13 to 0.17], Standard Error of Mean 0.090

8. Secondary Outcome: Transition Dyspnea Index (TDI) at End of Treatment (Day 28)
Description: TDI measures changes in dyspnea severity from the baseline as established by the Baseline Dyspnea Index (BDI). TDI is an interviewer-administered rating of severity of dyspnea that assesses Change in Functional Impairment, Change in Magnitude of Task, and Change in Magnitude of Effort domains on a 7-point scale ranging from -3 (major deterioration) to +3 (major improvement). Total score ranges from -9 to +9. The lower the score, the more deterioration in severity of dyspnea.
Time Frame: Baseline to end of treatment (Day 28)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale | -1 (0.5) | -0 (0.5)
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; The ANCOVA model used TDI as the response variable with treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection and BDI as covariates; Test type: Superiority or Other; p = 0.433, ANCOVA; LS mean difference = -1, 90% CI 2-sided [-1.6 to 0.6], Standard Error of Mean 0.7

9. Secondary Outcome: Change From Baseline for the Morning PEF and Evening PEF of the Bronkotest Diary Card
Description: The Bronkotest diary card is a paper based diary card that was filled out by patients daily, recording values from morning and evening peak expiratory flow (PEF) measurements and answering 8 questions on signs and symptoms. Summary statistics for baseline (mean of the last 7 days prior to first dose) and change (mean of the last 7 days on treatment - baseline) only contain patients included in the analysis. For symptom scores a decrease is an improvement, for PEF an increase is an improvement.
Time Frame: Baseline and Last 7 days on treatment
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 26 | 25
L/min
  Morning PEF | -5.3 (5.41) | -5.9 (5.53)
  Evening PEF | -7.3 (4.95) | -10.6 (5.06)
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; Morning PEF: Analysis of covariance includes treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection and baseline as covariates; Test type: Superiority or Other; p = 0.935, ANCOVA; LS mean difference = 0.7, 90% CI 2-sided [-12.81 to 14.13], Standard Error of Mean 8.03
Statistical Analysis 2: Comparison: AZD5069 vs Placebo; Evening PEF: Analysis of covariance included treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection and baseline as covariates; Test type: Superiority or Other; p = 0.654, ANCOVA; LS mean difference = 3.3, 90% CI 2-sided [-9.02 to 15.64], Standard Error of Mean 7.35

10. Secondary Outcome: Change From Baseline for the Symptom Scores of the Bronkotest Diary Card
Description: The Bronkotest diary card is a paper based diary card that was filled out by patients daily, recording values from morning and evening peak expiratory flow (PEF) measurements and answering 8 questions on signs and symptoms. Symptom scores were recorded for night-time symptoms, breathing, sputum colour, sputum amount, sputum type, wellbeing, number of puffs of inhalers, and cough, generally scored on a scale from 0 (no symptoms) to 4 (worst symptoms). Summary statistics for baseline (mean of the last 7 days prior to first dose) and change (mean of the last 7 days on treatment - baseline) only contain patients included in the analysis. For symptom scores a decrease is an improvement, for PEF an increase is an improvement.
Time Frame: Baseline and Last 7 days on treatment
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale
  Describe your breathing | 0.1 (0.10) | -0.1 (0.10)
  How often do you cough? | 0.1 (0.09) | 0.0 (0.09)
  Night time symptom score | 0.4 (0.12) | 0.1 (0.12)
  What color is your sputum? | -0.7 (0.18) | -0.3 (0.18)
  The amount of sputum you produced | 0.1 (0.08) | 0.0 (0.09)
  Type of sputum | -0.3 (0.09) | -0.1 (0.09)
  How do you feel? | 0.2 (0.10) | -0.0 (0.10)
  Number of puffs of inhalers | 0.1 (0.30) | 0.2 (0.30)
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; Describe your breathing: Analysis of covariance included treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection and baseline as covariates; Test type: Superiority or Other; p = 0.329, ANCOVA; LS mean difference = 0.1, 90% CI 2-sided [-0.09 to 0.36], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: AZD5069 vs Placebo; How often do you cough?: Analysis of covariance included treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection and baseline as covariates; Test type: Superiority or Other; p = 0.664, ANCOVA; LS mean difference = 0.1, 90% CI 2-sided [-0.16 to 0.27], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: AZD5069 vs Placebo; Night time symptom score: Analysis of covariance includes treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection and baseline as covariates; Test type: Superiority or Other; p = 0.152, ANCOVA; LS mean difference = 0.3, 90% CI 2-sided [-0.04 to 0.54], Standard Error of Mean 0.17
Statistical Analysis 4: Comparison: AZD5069 vs Placebo; What color is your sputum?: Analysis of covariance included treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection and baseline as covariates; Test type: Superiority or Other; p = 0.150, ANCOVA; LS mean difference = -0.4, 90% CI 2-sided [-0.80 to 0.05], Standard Error of Mean 0.25
Statistical Analysis 5: Comparison: AZD5069 vs Placebo; The amount of sputum you produced: Analysis of covariance included treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection and baseline as covariates; Test type: Superiority or Other; p = 0.248, ANCOVA; LS mean difference = 0.1, 90% CI 2-sided [-0.06 to 0.35], Standard Error of Mean 0.12
Statistical Analysis 6: Comparison: AZD5069 vs Placebo; Type of sputum: Analysis of covariance included treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection and baseline as covariates; Test type: Superiority or Other; p = 0.053, ANCOVA; LS mean difference = -0.2, 90% CI 2-sided [-0.45 to -0.04], Standard Error of Mean 0.12
Statistical Analysis 7: Comparison: AZD5069 vs Placebo; How do you feel?: Analysis of covariance includes treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection and baseline as covariates; Test type: Superiority or Other; p = 0.179, ANCOVA; LS mean difference = 0.2, 90% CI 2-sided [-0.04 to 0.42], Standard Error of Mean 0.14
Statistical Analysis 8: Comparison: AZD5069 vs Placebo; Number of puffs of inhalers: Analysis of covariance includes treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection and baseline as covariates; Test type: Superiority or Other; p = 0.942, ANCOVA; LS mean difference = -0.0, 90% CI 2-sided [-0.75 to 0.68], Standard Error of Mean 0.43

11. Secondary Outcome: Change From Baseline Total and Domain Scores in St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C)
Description: SGRQ-C total score shows the impact of COPD on patient's health status, and expressed as a percentage of impairment with scale from 0 (best health status) to 100 (worst possible status). The SGRQ-C contains 3 domains:
  Symptom (distress due to respiratory symptoms), Activity (disturbance of physical activity) and Impact (overall impact on daily life and well being). All three domains with scale from 0 (best health status) to 100 (worst possible status).
Time Frame: Baseline and end of treatment (Day 28)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 25 | 26
units on a scale
  Total score | -1.75 (2.402) | -0.09 (2.355)
  Symptom domain | -3.16 (2.356) | 1.72 (2.309)
  Activity domain | -0.46 (3.216) | 0.85 (3.153)
  Impact domain | -1.83 (2.742) | -1.45 (2.689)
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; Total score: Analysis of covariance included treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection and baseline as covariates; Test type: Superiority or Other; p = 0.625, ANCOVA; LS mean difference = -1.66, 90% CI 2-sided [-7.32 to 4.00], Standard Error of Mean 3.374
Statistical Analysis 2: Comparison: AZD5069 vs Placebo; Symptom domain: Analysis of covariance included treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection and baseline as covariates; Test type: Superiority or Other; p = 0.151, ANCOVA; LS mean difference = -4.88, 90% CI 2-sided [-10.49 to 0.74], Standard Error of Mean 3.342
Statistical Analysis 3: Comparison: AZD5069 vs Placebo; Activity domain: Analysis of covariance included treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection and baseline as covariates; Test type: Superiority or Other; p = 0.773, ANCOVA; LS mean difference = -1.31, 90% CI 2-sided [-8.91 to 6.28], Standard Error of Mean 4.524
Statistical Analysis 4: Comparison: AZD5069 vs Placebo; Impact domain: Analysis of covariance included treatment, inhaled corticosteroids, Pseudomonas aeruginosa infection and baseline as covariates; Test type: Superiority or Other; p = 0.920, ANCOVA; LS mean difference = -0.39, 90% CI 2-sided [-6.84 to 6.07], Standard Error of Mean 3.845

12. Secondary Outcome: Ratio of Interleukin-1 Beta (IL-1β) in Sputum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 22 | 25
ratio | 0.63 [0.44 to 0.90] | 0.91 [0.65 to 1.28]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.220, ANCOVA; Ratio of LS means = 0.69, 90% CI 2-sided [0.42 to 1.14]

13. Secondary Outcome: Ratio of Interleukin-6 (IL-6) in Sputum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 22 | 25
ratio | 3.68 [2.79 to 4.84] | 0.82 [0.64 to 1.07]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Ratio of LS means = 4.46, 90% CI 2-sided [3.05 to 6.54]

14. Secondary Outcome: Ratio of Regulated on Activation, Normal T Cell Expressed and Secreted (RANTES) in Sputum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 22 | 25
ratio | 0.99 [0.79 to 1.24] | 1.07 [0.87 to 1.32]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.670, ANCOVA; Ratio of LS means = 0.92, 90% CI 2-sided [0.68 to 1.26]

15. Secondary Outcome: Ratio of Monocyte Chemoattractant Protein-1 (MCP-1) in Sputum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 22 | 25
ratio | 0.91 [0.77 to 1.09] | 0.92 [0.78 to 1.08]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.968, ANCOVA; Ratio of LS means = 0.99, 90% CI 2-sided [0.78 to 1.27]

16. Secondary Outcome: Ratio of Tumor Necrosis Factor Alpha (TNF-α) in Sputum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 22 | 25
ratio | 1.29 [0.93 to 1.80] | 0.91 [0.67 to 1.23]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.193, ANCOVA; Ratio of LS means = 1.43, 90% CI 2-sided [0.91 to 2.24]

17. Secondary Outcome: Ratio of Growth-related Oncogene-α (GRO-α) in Sputum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 22 | 25
ratio | 2.77 [2.08 to 3.67] | 0.85 [0.65 to 1.11]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Ratio of LS means = 3.24, 90% CI 2-sided [2.19 to 4.79]

18. Secondary Outcome: Ratio of Interleukin-8 (IL-8) in Sputum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 22 | 26
ratio | 0.81 [0.62 to 1.07] | 0.80 [0.62 to 1.02]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.917, ANCOVA; Ratio of LS means = 1.02, 90% CI 2-sided [0.71 to 1.48]

19. Secondary Outcome: Ratio of Neutrophil Elastase Activity in Sputum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 4 | 5
ratio | 0.34 [0.09 to 1.28] | 1.95 [0.59 to 6.39]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.111, ANCOVA; Ratio of LS means = 0.17, 90% CI 2-sided [0.03 to 1.08]

20. Secondary Outcome: Ratio of Serum Amyloid A (SAA) in Serum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 24 | 24
ratio | 1.18 [0.82 to 1.72] | 0.89 [0.61 to 1.29]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.367, ANCOVA; Ratio of LS means = 1.33, 90% CI 2-sided [0.79 to 2.26]

21. Secondary Outcome: Ratio of C-reactive Protein (CRP) in Serum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 24 | 24
ratio | 1.28 [0.94 to 1.76] | 0.83 [0.61 to 1.14]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.112, ANCOVA; Ratio of LS means = 1.54, 90% CI 2-sided [0.98 to 2.40]

22. Secondary Outcome: Ratio of Tumor Necrosis Factor Alpha (TNF-α) in Serum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 24 | 24
ratio | 1.02 [0.97 to 1.06] | 0.97 [0.92 to 1.02]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.241, ANCOVA; Ratio of LS means = 1.05, 90% CI 2-sided [0.98 to 1.12]

23. Secondary Outcome: Ratio of Growth-related Oncogene-α (GRO-α) in Serum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 16 | 24
ratio | 5.45 [4.42 to 6.73] | 0.99 [0.84 to 1.18]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Ratio of LS means = 5.50, 90% CI 2-sided [4.18 to 7.23]

24. Secondary Outcome: Ratio of Interleukin-6 (IL-6) in Serum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 24 | 24
ratio | 1.13 [0.96 to 1.34] | 0.97 [0.82 to 1.15]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.281, ANCOVA; Ratio of LS means = 1.16, 90% CI 2-sided [0.92 to 1.47]

25. Secondary Outcome: Ratio of Interleukin-1 Beta (IL-1β) in Serum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 24 | 24
ratio | 1.45 [1.25 to 1.67] | 0.93 [0.80 to 1.07]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.001, ANCOVA; Ratio of LS means = 1.56, 90% CI 2-sided [1.28 to 1.91]

26. Secondary Outcome: Ratio of Interleukin-8 (IL-8) in Serum at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits.
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | AZD5069 | Placebo
Number analyzed (Participants) | 24 | 24
ratio | 5.90 [4.74 to 7.34] | 0.97 [0.78 to 1.21]
Statistical Analysis 1: Comparison: AZD5069 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Ratio of LS means = 6.07, 90% CI 2-sided [4.42 to 8.35]

ADVERSE EVENTS:
Groups:
- AZD5069: 80 mg bd
- Placebo: Placebo for AZD5069 bd
Arm/Group | AZD5069 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/26
Other Adverse Events (participants affected / at risk) | 22/26 | 16/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD5069 (N=26) | Placebo (N=26)
Infective Exacerbation Of Bronchiectasis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD5069 (N=26) | Placebo (N=26)
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 2
Nasopharyngitis (Infections and infestations) | 3 | 5
Infective Exacerbation Of Bronchiectasis (Infections and infestations) | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 5 | 3
Somnolence (Nervous system disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days